CLINICAL TRIAL: NCT06097975
Title: A Phase I Clinical Trial on Combined (Neo-)Adjuvant Intravenous Plus Intracranial Administration of Ipilimumab and Nivolumab in Recurrent Glioblastoma
Brief Title: A Clinical Trial on Combined (Neo-)Adjuvant Intravenous Plus Intracranial Administration of Ipilimumab and Nivolumab in Recurrent Glioblastoma
Acronym: NEO-GLITIPNI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Bart Neyns, prof. dr., Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-BN-001
Record Dates: First submitted 2023-10-05; First posted 2023-10-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Neurosurgical Procedures; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Drug: Neo-adjuvant nivolumab and ipililumab IV + adjuvant nivolumab and ipililumab IV; Procedure: Neurosurgery and intracavitary injection nivolumab and ipililumab; Drug: Adjuvant nivolumab IV + nivolumab and ipililumab intracavitary

INTERVENTIONS:
Drug: Neo-adjuvant nivolumab and ipililumab IV + adjuvant nivolumab and ipililumab IV — Participants will receive neo-adjuvant administration of intravenous immunotherapy on day 1 + day 22: ipilimumab + nivolumab IV.
Procedure: Neurosurgery and intracavitary injection nivolumab and ipililumab — The neo-adjuvant therapy will be followed by a maximal safe surgery resection of the glioblastoma. Immunotherapy (nivolumab + ipililumab) will be injected into the brain tissue, followed by insertion of an Ommaya reservoir
Drug: Adjuvant nivolumab IV + nivolumab and ipililumab intracavitary — Postoperatively, administration of immunotherapy will be continued, on day 15 postoperatively and every 2 weeks thereafter patients will receive nivolumab IV as well as ipililumab + nivolumab intracavitary.

SUMMARY:
The goal of this phase I interventional study is to determine the safety and feasibility of the proposed investigational (neo-)adjuvant treatment regimen in patients with resectable reccurent glioblastoma.

Participants will:

* receive neo-adjuvant administration of intravenous immunotherapy
* followed by a maximal safe neurosurgical resection
* afterwards, immunotherapy will be injected into the brain tissue
* followed by insertion of an Ommaya reservoir
* postoperatively, administration of immunotherapy will be continued

ELIGIBILITY:
1. Subjects must have signed and dated an approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
2. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.
3. Histopathological diagnosis of glioblastoma (= IDHwt, WHO grade IV astrocytoma of the central nervous system (Louis, Perry et al. 2021).
4. Diagnosis of resectable glioblastoma recurrence and/or progression following prior standard of care treatment (surgery for resectable lesions, radiation therapy and temozolomide chemotherapy). Recurrence/progression is defined as significant [according to the investigators assessment] growth and/or recurrence of the glioblastoma tumor mass on sequential MRI of the brain;
5. The following disease characteristics should be present:

   1. Presence of a measurable tumor lesion that is characterized by gadolinium enhancement on T1-MRI of the brain (with a longest diameter of > 10 mm and a perpendicular diameter of >5mm).
   2. No evidence of clinically relevant spontaneous intra-tumor hemorrhage on baseline MRI-imaging or in the prior disease history;
6. No ventriculo-peritoneal drain:
7. No contraindication for evaluation by gadolinium enhanced MRI, 18FFET-PET/CT of the brain or whole-body contrast enhanced CT;
8. ECOG performance status score of 0, 1 or 2;
9. An interval of at least 4 months (: 16 weeks) after the end of postoperative radiation therapy for glioblastoma unless progression is confirmed on an MRI of the brain obtained > 4 week after the first observation of progression; and with an interval of at least 4 weeks after the last administration of temozolomide;
10. Male or female, 18 years of age or older;
11. Resolution of all acute treatment related adverse effects of prior surgical procedures, radiotherapy and temozolomide to NCI CTCAEv4.0 grade 0 or 1 except for alopecia;
12. Adequate organ function as defined by the following criteria:

    1. Total serum bilirubin < 1.5 x ULN (patients with Gilbert's disease exempt who should have bilirubin < 2x ULN)
    2. AST and ALT < 2.5 x upper limit of normal (ULN);
    3. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥60 mL/min
    4. Absolute neutrophil count (ANC) > 1500/mm³ without growth factor support
    5. Platelets > 75 000 cells/mm³
    6. Hemoglobin ≥9 g/dL (which may be obtained by transfusion or growth factor support)
    7. FT4 hormone levels within normal range;
13. No prior treatment on a nivolumab and/or ipilimumab trial;
14. No prior treatment with an anti-CTLA-4 or anti-PD-1/-L1 targeted therapy;
15. No gastrointestinal abnormalities including:

    1. Inability to take oral medication.
    2. Requirement for intravenous alimentation.
    3. Prior surgical procedures affecting absorption including gastric resection.
    4. Treatment for active peptic ulcer disease in the past 6 months.
    5. Malabsorption syndromes.
    6. Active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
16. No evidence of pre-existing uncontrolled hypertension as documented by baseline blood pressure reading. The baseline systolic blood pressure reading must be ≤140 mm Hg, and the baseline diastolic blood pressure readings must be ≤90 mm Hg. If baseline blood pressure reading exceeds the inclusion values a second blood pressure reading (taken at least 1 hour apart) must be documented in order to confirm the absence of uncontrolled hypertension. Patients whose hypertension is controlled by antihypertensive therapies are eligible;
17. No concurrent treatment:

    1. In another therapeutic clinical trial;
    2. No requirement for permanent therapeutic anticoagulation therapy.
18. Subjects with active, known, or suspected autoimmune disease are not eligible. Subjects with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll;
19. Subjects requiring systemic treatment with either corticosteroids (> 8 mg daily methylprednisolone equivalent) or other immunosuppressive medications within 14 days of study enrollment. Inhaled or topical steroids are permitted in the absence of active autoimmune disease;
20. No active uncontrolled seizure disorder;
21. No myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure or any unstable arrhythmia, cerebrovascular accident or transient ischemic attack, within the 12 months prior to study drug administration.;
22. No known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness;
23. No serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment;
24. No history of a malignancy (other than glioma) except those treated with curative intent for skin cancer (other than melanoma) or in situ breast or cervical cancer or those treated with curative intent for any other cancer with no evidence of disease for 5 years;
25. No other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study;
26. No dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol;
27. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception measures during the period of therapy, which should be continued for at least 5 months following the last dose of nivolumab as indicated in the SmPC. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment and pregnancy testing should be conducted within 24h prior to the first dose of immune checkpoint inhibitors and thereafter monthly and at the end of systemic exposure. The definition of effective contraception will be included in the Informed consent form. Women must not be breastfeeding at initiation of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and feasibility of the proposed investigational (neo-)adjuvant treatment regimen in patients with resectable recurrent glioblastoma. | 1 year
  Incidence of treatment related adverse events (TRAE). TRAE will be collected on a continuous basis. Type, frequency and severity (graded according to the CTCAEv5) will be reported descriptively.

SECONDARY OUTCOMES:
Estimate anti-tumor responses of the proposed investigational (neo-)adjuvant treatment regimen. | 4 years
  Objective response rate (ORR, according to iRANO criteria) following 4 weeks of neo-adjuvant therapy.

OTHER OUTCOMES:
Estimate progression-free and overall survival estimated by Kaplan-Meier survival estimates. | 4 years
  PFS and OS estimated by Kaplan-Meier survival analysis (incl. median, 6-months-, and yearly survival rates with 95% CI).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No